CLINICAL TRIAL: NCT04890301
Title: Puncture Template Assisted CT Guided Versus Simple CT Guided Biopsy for Small Pulmonary Nodules: a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Puncture Template Assisted Biopsy for Pulmonary Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNRBG-2021-PT-PN
Record Dates: First submitted 2021-04-30; First posted 2021-05-18 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Nodule; CT Guided Biopsy
Keywords: pulmonary nodule; biopsy; puncture template

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puncture Template and CT group (Experimental): Puncture Template assisted CT guided lung biopsy was performed.
  Interventions: Behavioral: CT guided biopsy for pulmonary nodule
- CT group (Active Comparator): Simple CT guided lung biopsy was performed.
  Interventions: Behavioral: CT guided biopsy for pulmonary nodule

INTERVENTIONS:
Behavioral: CT guided biopsy for pulmonary nodule — The technical process of the experimental group: ① design of puncture path, positioning and fixation of patients; ② puncture point positioning; ③ installation of navigation frame and template; ④ percutaneous lung biopsy guided by PT combined with CT.
  The technical process of the active comparator group: ① planning puncture path, positioning and fixation of patients; ② positioning puncture point; ③ CT guided percutaneous lung biopsy.
  The operation related information, complications and postoperative pathological results were collected.

SUMMARY:
Pulmonary nodules are small in size and easy to move with breathing. CT guided puncture is highly dependent on the personal experience of physicians, that is, the accuracy, efficiency and incidence of complications of puncture vary greatly among physicians.

Puncture template (PT) assisted CT guided needle biopsy of pulmonary nodules has good clinical feasibility, which is expected to make up for the deficiency of simple CT guided needle biopsy, and make the needle biopsy of pulmonary nodules more accurate and standardized.

This study intends to carry out a randomized controlled study to further evaluate the safety and effectiveness of PT assisted CT guided needle biopsy of pulmonary nodules, and provide higher quality data reference for its clinical application.

Patients were randomly divided into two groups: PT assisted CT guided or simple CT guided lung biopsy. The operation related information, complications and postoperative pathological results of the two groups were collected.

Primary end point: puncture accuracy Secondary end point: success rate of first needle puncture; complication rate (such as pneumothorax, bleeding, etc.); operation time; CT scan times; pathologic findings.

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple pulmonary nodules (solid, partially solid, pure ground glass), with the maximum diameter of 5mm to 20mm and need for pathological diagnosis.
* No drugs affecting blood coagulation and (or) platelet aggregation were used; if used, the drugs had been stopped for enough time according to the drug elution period.
* KPS > 60, no serious or uncontrollable underlying diseases, the patients can tolerate lung puncture according to clinical evaluation.
* There is an appropriate puncture path.

Exclusion Criteria:

* Poor lung function (such as FEV1 < 40% in the first second and / or DLCO < 50%) and / or isolated pulmonary bullae on the puncture path.
* The nodule is close to small airway and blood vessels, or has pulmonary hypertension and superior vena cava compression, so the risk of puncture bleeding and hemoptysis is expected to be high.
* Poor compliance, unable to complete the cooperation.
* Due to other reasons which is not suitable to participate in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Puncture accuracy assessed by direct measurement. | Immediately after the operation (puncture).
  The distance between the actual puncture point and the expected puncture point should be measured on CT image, to get whether there are any errors in the needle insertion of the two groups and whether there are differences between the two groups.

SECONDARY OUTCOMES:
Success rate of first needle puncture assessed by freqencey of needle adjustment. | Immediately after the operation (puncture).
  The freqencey of times of needle adjustment should be recorded. If the frequency of puncture needle adjustment is 0, the first needle puncture was recorded as successful. If the frequency of needle adjustment is not 0, the number of times of needle adjustment should be recorded.
Complications assessed by CTCAE 5.0 | From the beginning of operation to 1 month after operation (puncture).
  The incidence and severity of complications such as pneumothorax, subcutaneous emphysema, hemothorax, hemoptysis and air embolism should be recorded.
Operation time assessed by direct timing. | Immediately after the operation (puncture).
  The time from the first CT scan to the last CT scan should be recorded.
Times of CT scans assessed by direct counting. | Immediately after the operation (puncture).
  The total number of CT scans throughout the operation should be recorded.
Pathological report issued by pathology department. | 1 week to 1 month after operation (puncture).
  The pathological results (pathological report issued by pathology department) of puncture should be followed up and recorded. If the pathological results indicate normal tissue/structure, the puncture result is considered to be negative.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, Principal Investigator — Peking University Third Hospital, Department of Radiation Oncology
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other researchers and can be requested by the email of study sponsor.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available within 2 years of the study completion.
Access Criteria: The purpose needs to be informed to and judged by the research sponsor. Requestors will be required to sign a Data Access Agreement.